CLINICAL TRIAL: NCT03521596
Title: Non-invasive Diagnostics and Monitoring of Minimal Residual Disease and Clonal Evolution in Waldenström's Macroglobulinemia and in IgM Monoclonal Gammopathy of Undetermined Significance
Brief Title: Non-invasive Diagnostics and Monitoring of MRD and Clonal Evolution in Waldenström's Macroglobulinemia and in IgM-MGUS
Acronym: FIL_BIOWM
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_BIOWM
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: IgM monoclonal gammopathy; Waldenström's Macroglobulinemia; Minimal residual disease; Clonal evolution
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Neoplasm, Residual | interventions — Clonal Evolution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Peripheral blood, Bone marrow and Urine collected at Baseline, Before treatment, after treatment, at 12 months follow up, at 24 months follow up and at 60 months follow up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient enrolled: Part of the patients will be retrospectively enrolled (learning sample) and part prospectively (validation sample)
  Interventions: Other: MRD and clonal evolution

INTERVENTIONS:
Other: MRD and clonal evolution — Patient evaluation at the time of diagnosis and during the disease course using highly sensitive techniques

SUMMARY:
Multicenter retrospective and prospective observational study including patients with WM or IgM-MGUS evaluated at the time of diagnosis and during the disease course using highly sensitive techniques.

DETAILED DESCRIPTION:
Multicenter retrospective and prospective observational study including patients with WM or IgM-MGUS evaluated at the time of diagnosis and during the disease course using highly sensitive techniques such as flow cytometry, real time quantitative PCR (RT-qPCR), digital droplet PCR (dd-PCR) and NGS, in order to: evaluate the mutational status on genomic DNA or cell-free DNA and compare the results to assess the most reliable source for mutation studies; perform and compare molecular and flow cytometry analyses on bone marrow, peripheral blood (both analyses), plasma and urine samples (only molecular analysis) to assess the best source for diagnosis and MRD monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IgM monoclonal gammopathy of undetermined significance (Ig-MGUS) or Waldenström's Macroglobulinemia (WM) according to criteria established at the second International Workshop on Waldenström's Macroglobulinemia [1]
* Age ≥ 18 years
* Previously untreated patients (only for the prospective cohort)
* Symptomatic or asymptomatic disease
* Subject understands and voluntarily signs an informed consent form approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB)

Exclusion Criteria:

* Active HBV, HCV or HIV infection (antiHBc+ patients with undetectable HBV-DNA are eligible to the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include either IgM-MGUS, asymptomatic WM or symptomatic WM patients requiring treatment. Patients in need of therapy will be treated according to recently published guidelines [49]. Patients treated with new agents, including the BTK inhibitor Ibrutinib, will be included. Patient enrolled retrospectively will constitute the learning cohort of the study, while those enrolled prospectively will constitute the validation cohort).
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Rate of mutation | 22 months
  To demonstrate that the rate of mutations of MYD88 (L265P) and/or CXCR4 (S338X) detected in peripheral blood and/or urine show a negligible difference with the rate of mutations detected in bone marrow samples (BM, gold standard)

CONTACTS AND LOCATIONS:
Overall Officials: Marzia Varettoni, Principal Investigator — Pavia - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia
Locations (14):
- Italy (14):
  - Divisione di Ematologia Ospedale Niguarda, Milan, MI
  - SOS Ematologia Ospedale C. Massaia, Asti
  - IRCCS Istituto Tumori Giovanni Paolo II - UOC Ematologia, Bari
  - AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - A.O. Universitaria Di Parma, Parma
  - Ematologia Policlinico San Matteo, Pavia
  - AO Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - Ospedale degli Infermi di Rimini, Rimini
  - Policlinico A. Gemelli Università Cattolica del Sacro Cuore, Roma
  - UOC Ematologia, AOU Senese, Siena
  - A.O. Città della Salute e della Scienza Ematologia Universitaria, Torino
  - Azienda Sanitaria Universitaria Integrata di Udine (A.S.U.I. Udine) - PO S. Maria della Misericordia, Udine
  - Ematologia - OSPEDALE DI CIRCOLO E FONDAZIONE MACCHI, Varese